CLINICAL TRIAL: NCT01660997
Title: MLN9708 and Dexamethasone in High Risk Smoldering Multiple Myeloma: A Clinical and Correlative Pilot Study
Brief Title: MLN9708 and Dexamethasone for High-Risk Smoldering Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120180; 12-C-0180
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-03-11

CONDITIONS: Multiple Myeloma
Keywords: Proteasome Inhibitor; Induction Combination Therapy; Maintenance Strategy; Potent Anti-Myeloma Effect; Precursor Disease
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Dexamethasone

INTERVENTIONS:
Drug: MLN9708
Drug: Dexamethasone

SUMMARY:
Background:

- Smoldering multiple myeloma (SMM) is a condition that can lead to multiple myeloma, a type of blood cancer. In many high-risk cases, SMM can develop into multiple myeloma in less than 2 years. The current standard of care for SMM is follow-up without treatment until multiple myeloma develops. However, some drugs are being studied to see if they can slow down or prevent the disease from progressing. One such drug is MLN9708. It has shown some results against multiple myeloma. Researchers want to combine MLN9708 with dexamethasone to see how it works against high-risk SMM.

Objectives:

- To see if MLN9708 with dexamethasone is a safe and effective treatment for high-risk smoldering multiple myeloma.

Eligibility:

- Individuals at least 18 years of age who have high-risk smoldering multiple myeloma.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies and a bone marrow biopsy may also be performed.
* Participants will take MLN9708 and dexamethasone on a regular schedule for 28 days. They will take each drug four times at regular intervals during each cycle of treatment.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Participants will have 12 cycles of treatment. After four cycles, patients will be recommended to have their own stem cells collected and stored. This will allow the potential application of a highdose melpahalan/autologous stem cell transplant in the event there is a need in the future (not part of this study).
* After 12 cycles, participants will keep taking MLN9708 as long as the disease does not progress and the side effects are not too severe.

DETAILED DESCRIPTION:
Background:

* SMM is a precursor condition to MM defined by the clinical parameters of M-protein greater than or equal to 3.0 g/dL or bone marrow plasma cells greater than or equal to 10% and absence of end organ disease.
* Risk of progression of high risk SMM at 5 years is 72-75% with median time to progression less than 2 years.
* The current standard of care for SMM is close follow-up without treatment until symptomatic MM develops. However, IMWG states Preventive clinical trials need to be considered for patients with high risk smoldering myeloma .
* MLN9708 is a new oral proteasome inhibitor with potent anti-MM effects

Objectives:

Primary Endpoint:

-The primary objective of the study is to assess the response rate of MLN9708/low-dose

dexamethasone in patients with high-risk SMM.

Secondary Endpoints:

* To determine progression free survival (PFS)
* To determine duration of response (DOR)
* To evaluate toxicity of combination therapy (MLN9708 and low-dose dexamethasone).
* To evaluate biological activity of MLN9708 and correlate to clinical outcomes (gene expression profiling and proteasome activity and ubiquination assays, and effects on downstream signaling targets using pre- and post-MLN9708 exposure bone marrow samples)

Eligibility:

* SMM according to the International Myeloma Working Group definition i.e.:

  * Serum M-protein greater than or equal to 3 g/dl and/or bone marrow plasma cells greater than or equal to 10 %,
  * Absence of anemia: Hemoglobin greater than10 g/dl
  * Absence of renal failure: calculated creatinine clearance (according to MDRD) greater than 80 ml/min (or alternatively based on standard creatinine level criteria of 2 mg/dl)
  * Absence of hypercalcemia: Ca < 10.5 mg/dl or less than or equal to 2.5 mmol/L
  * Absence of lytic bone lesion
* Measurable disease within the past 4 weeks defined by any one of the following:

  * Serum monoclonal protein greater than or equal to 1.0 g/dl
  * Urine monoclonal protein >200 mg/24 hour
  * Serum immunoglobulin free light chain >10 mg/dL AND abnormal kappa/lambda ratio (reference 0.26-1.65)
* High-risk SMM per Mayo Clinic or Spanish PETHEMA criteria
* Age greater than18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Ability to give informed consent
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than1.0 K/uL
  * platelets greater than75 K/uL (Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrolment.)
  * hemoglobin greater than 8 g/dL(transfusions are permissible)
  * total bilirubin less than1.5 X institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) less than 3.0 X institutional upper limit of normal

Design:

-Single arm pilot trial of combination therapy (MLN9708 and dexamethasone) for high risk smoldering multiple myeloma

* Patients will receive 12 cycles (28 days each) of induction combination therapy of MLN9708 and low-dose dexamethasone. After 12 cycles of MLN9708/low-dose dexamethasone, patients will receive MLN9708 maintenance until progression or unacceptable toxicity.
* Patients will have routine blood work with SPEP and free light chains monthly
* Pre- and post-treatment bone marrow biopsies will be obtained for confirmation of diagnosis and correlative studies
* Patients will also undergo evaluation for minimal residual disease at complete remission/completion of 12 cycles of therapy, using multi-parametric flow cytometry and FDG PET-CT
* This single arm pilot study will enroll 12 evaluable patients and determine M-spike levels on each patient immediately pre-treatment as well as after completing 12 cycles of treatment. The study aim is to find 9 or more patients (out of 12) with a partial response (PR) or better; which would provide strong evidence that the true probability of an overall response is consistent with 80% or more.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed Smoldering Multiple Myeloma confirmed by the Laboratory of Pathology, NCI based on the International Myeloma Working Group Criteria:

  * Serum M-protein greater than or equal to 3 g/dl and/or bone marrow plasma cells greater than or equal to 10 %,
  * Absence of anemia: Hemoglobin >10 g/dl
  * Absence of renal failure: calculated creatinine clearance (according to MDRD) > 80 ml/min (or alternatively based on standard creatinine level criteria of 2 mg/dl)
  * Absence of hypercalcemia: Ca < 10.5 mg/dl or less than or equal to 2.5 mmol/L
  * Absence of lytic bone lesion
* High-risk SMM per Mayo Clinic2 or Spanish PETHEMA1 criteria
* Measurable disease within the past 4 weeks defined by any one of the following:

  * Serum monoclonal protein greater than or equal to 1.0 g/dl
  * Urine monoclonal protein >200 mg/24 hour
  * Serum immunoglobulin free light chain >10 mg/dL AND abnormal kappa/lambda ratio (reference 0.26-1.65)
* Age >18 years.
* ECOG performance status <2.
* Ability to give informed consent.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count >1.0 K/uL
  * Platelets >75 K/uL (Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.)
  * hemoglobin > 8 g/dL(transfusions are permissible)
  * total bilirubin <1.5 X institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) < 3.0 X institutional upper limit of normal
* Female patients who:

  * Are postmenopausal for at least 1 year before the Screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study treatment, OR agree to completely abstain from heterosexual intercourse.

    * The 2 methods of reliable contraception must include 1 highly effective method and 1 additional effective (barrier) method. Females of childbearing potential must be referred to a qualified provider of contraceptive methods if needed. The following are examples of highly effective and additional effective methods of contraception:
* Highly effective methods:

  * Intrauterine device (IUD)
  * Hormonal (birth control pills, injections, implants)
  * Tubal Ligation
  * Partner's Vasectomy

Additional effective methods:

* Male condom
* Diaphragm
* Cervical Cap

  -Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:
* Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study treatment, OR agree to completely abstain from heterosexual intercourse.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents not included in this trial, within 21 days of the start of this trial and throughout the duration of this trial.
* Prior therapy for SMM with a proteasome inhibitor.
* Patients with a diagnosis of MM.
* Contraindication to any concomitant medication, including antivirals, anticoagulation prophylaxis, tumor lysis prophylaxis, or hydration given prior to therapy.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Uncontrolled hypertension or diabetes.
* Pregnant or lactating females.
* Has refractory GI disease with refractory nausea/vomiting, inflammatory bowel disease, or bowel resection that would prevent absorption.
* Patient has greater than or equal to Grade 2 peripheral neuropathy.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Systemic treatment, within 14 days before study enrollment, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John s wort.
* Ongoing or active systemic infection, known human immunodeficiency virus (HIV) positive, known active hepatitis B virus hepatitis, or known active hepatitis C virus hepatitis.
* Co-morbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Psychiatric illness/social situation that would limit compliance with study requirements.
* QTc > 470 milliseconds (msec) on a 12-lead EKG obtained during the Screening period. If a machine reading is above this value, the EKG should be reviewed by a qualified reader and confirmed on a subsequent EKG.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements or GI procedure that could interfere with the oral absorption or tolerance of treatment.
* Major surgery within 1 month prior to enrollment.
* Radiotherapy within 14 days before enrollment.
* Central nervous system involvement (based on clinical assessment).
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
* No current bisphosphonate therapy (However, prior bisphosphonates or once a year intravenous bisphosphonate for osteoporosis is allowed).
* Patients with Paget s disease of the bone
* Recruitment Strategies
* Patients from the SMM and MGUS Natural History Study (NCI Protocol: 10-C-0096) will be potential candidates.
* Other participant sources will be from outside physician referrals.
* Our ongoing natural history study and outside physician referral network have a high representation of minorities.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07-30; Primary Completion 2014-03-11 (Actual); Study Completion 2014-03-11 (Actual)

PRIMARY OUTCOMES:
Response rate | 3 years

SECONDARY OUTCOMES:
Progression-free survival | 4 years
Duration of response | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Carl O Landgren, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Perez-Persona E, Vidriales MB, Mateo G, Garcia-Sanz R, Mateos MV, de Coca AG, Galende J, Martin-Nunez G, Alonso JM, de Las Heras N, Hernandez JM, Martin A, Lopez-Berges C, Orfao A, San Miguel JF. New criteria to identify risk of progression in monoclonal gammopathy of uncertain significance and smoldering multiple myeloma based on multiparameter flow cytometry analysis of bone marrow plasma cells. Blood. 2007 Oct 1;110(7):2586-92. doi: 10.1182/blood-2007-05-088443. Epub 2007 Jun 18. PMID 17576818
- [Background] Dispenzieri A, Kyle RA, Katzmann JA, Therneau TM, Larson D, Benson J, Clark RJ, Melton LJ 3rd, Gertz MA, Kumar SK, Fonseca R, Jelinek DF, Rajkumar SV. Immunoglobulin free light chain ratio is an independent risk factor for progression of smoldering (asymptomatic) multiple myeloma. Blood. 2008 Jan 15;111(2):785-9. doi: 10.1182/blood-2007-08-108357. Epub 2007 Oct 17. PMID 17942755
- [Background] Kyle RA, Durie BG, Rajkumar SV, Landgren O, Blade J, Merlini G, Kroger N, Einsele H, Vesole DH, Dimopoulos M, San Miguel J, Avet-Loiseau H, Hajek R, Chen WM, Anderson KC, Ludwig H, Sonneveld P, Pavlovsky S, Palumbo A, Richardson PG, Barlogie B, Greipp P, Vescio R, Turesson I, Westin J, Boccadoro M; International Myeloma Working Group. Monoclonal gammopathy of undetermined significance (MGUS) and smoldering (asymptomatic) multiple myeloma: IMWG consensus perspectives risk factors for progression and guidelines for monitoring and management. Leukemia. 2010 Jun;24(6):1121-7. doi: 10.1038/leu.2010.60. Epub 2010 Apr 22. PMID 20410922